CLINICAL TRIAL: NCT00279773
Title: A Phase I Dose Escalating Study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamics of TKI258 in Subjects With Acute Myeloid Leukemia
Brief Title: Safety, Pharmacokinetics and Pharmacodynamics of TKI258 in Subjects With Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study was stopped due to time dependent drug accumulation
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTKI258A2102
Record Dates: First submitted 2006-01-18; First posted 2006-01-20 (Estimated); Last update posted 2010-06-30 (Estimated); Status verified 2010-06

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute; Myeloid; Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

ARMS (2):
- TKI258 - dose escalation (Experimental): Dose-Escalation
  Interventions: Drug: TKI258
- TKI258 - dose expansion (Experimental): Dose-Expansion
  Interventions: Drug: TKI258

INTERVENTIONS:
Drug: TKI258

SUMMARY:
The primary objective is to determine the maximum tolerated dose (MTD), dose limiting toxicity (DLT), and safety profile of TKI258 when administered to subjects with acute myeloid leukemia (AML).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Acute Myeloid Leukemia
* Eighteen years of age or older
* Life expectancy of at least 2 months

Exclusion Criteria:

* Intracranial disease or epidural disease
* Clinically significant cardiac disease
* Diabetes mellitus uncontrolled with medication
* Pregnant or breast feeding women
* Dementia or altered mental status
* Known pre-existing clinically significant or uncontrolled disorder of the hypothalamic-pituitary axis, adrenal or thyroid glands
* Previous pericarditis
* Malabsorption syndrome or uncontrolled gastrointestinal symptoms such as nausea,diarrhea,vomiting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2004-09; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 28 days - dose-escalation; 4 months - dose-expansion
Dose limiting toxicity | 28 days - dose-escalation; 4 months - dose-expansion
Safety profile | 28 days - dose-escalation; 4 months - dose-expansion

SECONDARY OUTCOMES:
Evaluation of plasma pharmacokinetics and pharmacodynamics | 28 days - dose-escalation; 4 months - dose-expansion

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- The University of Texas, M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Wang X, Kay A, Anak O, Angevin E, Escudier B, Zhou W, Feng Y, Dugan M, Schran H. Population pharmacokinetic/pharmacodynamic modeling to assist dosing schedule selection for dovitinib. J Clin Pharmacol. 2013 Jan;53(1):14-20. doi: 10.1177/0091270011433330. Epub 2013 Jan 24. PMID 23400739